CLINICAL TRIAL: NCT01191814
Title: A Randomized Trial Comparing Covered Metal and Plastic Stents for Preoperative Biliary Decompression in Pancreatic Cancer
Brief Title: Comparison of Metal and Plastic Stents for Preoperative Biliary Decompression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Collaborators: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FT356090
Record Dates: First submitted 2010-08-12; First posted 2010-08-31 (Estimated); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Obstructive Jaundice; Pancreatic Cancer
Keywords: pancreatic cancer; obstructive jaundice; Obstructive jaundice secondary to pancreatic cancer
MeSH Terms: conditions — Jaundice, Obstructive; Pancreatic Neoplasms | interventions — Self Expandable Metallic Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metal stent (Active Comparator): Patients with pancreatic cancer causing bile duct obstruction will be treated by placement of a metal stent.
  Interventions: Procedure: Metal stent
- Plastic Stent (Active Comparator): Patients with pancreatic cancer causing bile duct obstruction will be treated by placement of a plastic stent
  Interventions: Procedure: Plastic stent

INTERVENTIONS:
Procedure: Metal stent — Patients with pancreatic cancer causing bile duct obstruction will be treated by placement of a metal stent.
  Arms: Metal stent
Procedure: Plastic stent — Patients with pancreatic cancer causing bile duct obstruction will be treated by placement of a 10Fr plastic stent.
  Arms: Plastic Stent

SUMMARY:
Covered self expandable metal stents (CSEMS) are three times larger in diameter than 10 Fr plastic stents. When compared to plastic stents, randomized trials have shown longer patency and fewer stent-related complications for CSEMS. The investigators hypothesize that placement of CSEMS would be a better treatment option for preoperative biliary decompression in patients with pancreatic cancer.

DETAILED DESCRIPTION:
Covered self expandable metal stents (CSEMS) are three times larger in diameter than 10 Fr plastic stents. When compared to plastic stents, randomized trials have shown longer patency and fewer stent-related complications for CSEMS. The investigators hypothesize that placement of CSEMS would be a better treatment option for preoperative biliary decompression in patients with pancreatic cancer as there will be better drainage of the obstructed biliary system with fewer adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pancreatic cancer and mass in the head of pancreas causing jaundice.
* Patients 19 yrs of age and older
* Serum bilirubin > 2mg/dl
* CT: No evidence of distant metastasis or local vascular invasion (tumor surrounding portal or mesenteric vessels for more than 180 degrees of their circumference or an irregular vessel margin).

Exclusion Criteria:

* Karnofsky score < 60
* Prior (ERCP or PTC) attempts at biliary decompression for the same indication
* Tumor-related gastric outlet obstruction (vomiting and oral intake of < 1L/day)
* Ongoing or planned neoadjuvant therapy
* Cholangitis at presentation or coagulopathy needing reversal medication
* Post-surgical anatomy
* Multiple extra-hepatic biliary strictures or concomitant stricture in liver hilum
* Failed ERCP's (Definition: Inability to deploy a biliary stent thereby requiring a PTC or surgery).

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-07; Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
Complications related to stent dysfunction | 30 days
  Complications related to stent dysfunction which include hyperbilirubinemia or cholangitis that warrant stent exchange (repeat intervention by ERCP)

SECONDARY OUTCOMES:
Procedural complications | 30 days
  Complications related to the procedure which includes pancreatitis, perforation or hemorrhage.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hasan, MD, Principal Investigator — AdventHealth
Locations (1):
- AdventHealth, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No
A manuscript will be developed following the closure of the study.